CLINICAL TRIAL: NCT04052126
Title: An Interventional Prospective Study to Test the Feasibility of an Individualized Physical Activity Program in Patients Over 65 Years of Age With Hematologic Malignancies: the OCAPI Project.
Brief Title: An Individualized Physical Activity Program in Patients Over 65 Years With Hematologic Malignancies
Acronym: OCAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OCAPI
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Aged; Aged, 80 and Over; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Exercise; Quality of Life; Fatigue
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized physical activity program (Experimental)
  Interventions: Other: Individualized physical activity program

INTERVENTIONS:
Other: Individualized physical activity program — Participants who agreed to participate in the study will participate in an individualized 6-month physical activity (PA) program, consisting of 3 periods: initiation (1st month), transition (2nd-3rd months) and autonomy (4th-6th months). It is based on 4 PA modalities:
  The supervised PA session in a sterile room or at home once a week during the initiation and transition phases (20-45 min, low-to-moderate intensity, walking, muscle strengthening, balance and flexibility exercises).
  The unsupervised PA session in a sterile room or at home once a week during the transition phase and twice a week during the autonomy phase (same as supervised session).
  Follow-up by telephone once a month during the autonomy phase (30 min, support to PA).
  Continuously wearing an activity tracker throughout the entire program (promotion of walking).
  Activities are planned over a period of 6 months to achieve an intervention that meets the key principles of progression, specificity and empowerment.

SUMMARY:
Older people with cancer differ from younger patients due to the combined effects of aging, comorbidities and cancer treatments on their health. In acute myeloid leukemia (AML) and non-hodgkin lymphoma (NHL), chemotherapy, which is the main treatment, is associated with significant toxicity that negatively affects patients' physical capacities and quality of life, already declining with age and comorbidities. It therefore seems essential to develop and evaluate interventions that can prevent physical and psychosocial decline and its consequences in these populations. However, no studies have evaluated a physical activity (PA) program among these populations, although the absence of risk of implementing PA during intense therapeutic procedures has been confirmed.

OCAPI is an interdisciplinary, prospective, interventional, feasibility study. It is intended to include 20 AML and 20 NHL patients 65 years of age or older at the time of initiation of the first chemotherapy line, with an ECOG <3, with no contraindications to PA and no history or coexistence of other primary cancer.

Expected results are to demonstrate that a program offering supervised sessions in a sterile room or at home and remote support can enable patients with AML or NHL to perform their daily PA in autonomy. All these results will generate preliminary data before implementing a larger national study.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and over,
* With histologically confirmed non-Hodgkin's lymphoma (NHL) or acute myeloid leukemia (AML),
* Requiring a first line of chemotherapy treatment or Azacitidine - Vénétoclax combination,
* Followed-up in one of the investigating centers,
* Residing in one of the following departments: Ain, Ardèche, Drôme, Isère, Loire, Rhône, Savoie, Haute-Savoie,
* Having a ECOG < 3,
* With a life expectancy > 6 months,
* Whose ability to engage in physical activity has been certified by a medical certificate issued by the investigator physician,
* Available and willing to participate in the study for the duration of the intervention and follow-up,
* Able to understand, read and write French,
* Affiliated with a social security scheme,
* Having dated and signed an informed consent.

Exclusion Criteria:

* Personal history or co-existence of another primary cancer (except of in situ cancer regardless of the site and/or basal cell skin cancer and/or non-mammary cancer in complete remission for more than 5 years),
* Treated by immunotherapy alone,
* Participating in concurrent physical activity studies,
* Deprived of their liberty by court or administrative decision.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Compliance rate of the physical activity sessions | 6 months
  Ratio of the number of supervised and unsupervised sessions performed by patients / number of scheduled sessions
Compliance rate of the phone calls | 6 months
  Ratio of the number of phone calls performed / number of scheduled calls
Compliance rate of the activity tracker | 6 months
  Ratio of the number of days wearing the activity tracker / number of days of the program

SECONDARY OUTCOMES:
Acceptability of the intervention | At inclusion
  Ratio of number of patients included / number of eligible patients
Safety of the intervention | 6 months
  Number, type and timing of program-related adverse events
Adherence of the intervention | 3 months and 6 months
  Ratio of the number of patients still in the program / number of patients included in the study
Impact of the program on autonomy for activities of daily living | At inclusion, 3 months and 6 months
  Activities of Daily Living questionnaire (ADL) - scale from 0 to 6, 0=autonomy; 6 = no autonomy
Impact of the program on autonomy for instrumental activities of daily living | At inclusion, 3 months and 6 months
  Instrumental activities of Daily Living questionnaire (IADL) - scale from 0 to 4, 0=autonomy; 4 = no autonomy
Impact of the program on upper body strength | At inclusion, 3 months and 6 months
  30-s Arm Curl Test
Impact of the program on lower body strength | At inclusion, 3 months and 6 months
  30-s Chair Stand Test
Impact of the program on upper body flexibility | At inclusion, 3 months and 6 months
  Back Scratch Test
Impact of the program on lower body flexibility | At inclusion, 3 months and 6 months
  Chair Sit and Reach Test
Impact of the program on agility | At inclusion, 3 months and 6 months
  Timed Up and Go Test
Impact of the program on walking endurance | At inclusion, 3 months and 6 months
  6-min Walk Test
Impact of the program on walking speed | At inclusion, 3 months and 6 months
  10-m Walk Test
Impact of the program on balance | At inclusion, 3 months and 6 months
  Open-eyes Unipodal Test
Impact of the program on grip strength | At inclusion, 3 months and 6 months
  Hand Grip Dynamometer Test
Impact of the program on anthropometrics | At inclusion, 3 months and 6 months
  BMI (weight and height will be combined to report BMI in kg/m^2)
Impact of the program on nutrition | At inclusion, 3 months and 6 months
  Mini Nutritional Assessment (MNA) - scale from 0 to 30 points; score<17=bad nutritional status ; 17 and 23.5=risk of malnutrition ; >24: adaptednutritional status
Impact of the program on cognition | At inclusion, 3 months and 6 months
  Montreal Cognitive Assessment (MoCA) ; scale from 0 to 30; normal if score >16
Impact of the program on depression | At inclusion, 3 months and 6 months
  Geriatric Depression Scale-15 (GDS-15) ; scale from 0 to 15 ; 0 to 5=normal ; 6 and 9 = high probability of depression ; > 9 = almost systematic depression
Impact of the program on self-efficacy | At inclusion, 3 months and 6 months
  Self-efficacy for exercise scale - This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Impact of the program on comorbidities | At inclusion, 3 months and 6 months
  Cumulativ Illness Rating Scale - Geriatric (CIRS-G) ; 14 items ; for each one, score from 0 to 4 : 0=no problem and 4=serious issue
Impact of the program on health-related quality of life | At inclusion, 3 months, 6 months and 1 year
  European Organization for Research and Treatment of Cancer core quality of life questionnaire (EORTC QLQ-C30) - scale from 0 to 100
Impact of the program on fatigue | At inclusion, 3 months, 6 months and 1 year
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) ; score from 0 to 65 ; the higher the score is, the less the patient has fatigue
Impact of the program on the level of physical activity | At inclusion, 3 months, 6 months and 1 year
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) ; Godin scale score: < 14 units: insufficiently active/sedentary ; 14-23: moderately active ; 24 or more : active
Impact of the program on exercise barriers | At inclusion, 3 months, 6 months and 1 year
  Barriers to Being Active Quiz
Impact of the program on social vulnerability | At inclusion and 1 year
  Évaluation de la précarité et des inégalités de santé pour les CES (EPICES questionnaire) - scale from 0 to 100, 0= no social vulnerability, 100=max vulnerability, threshold=30
Impact of the program on falls | At inclusion and 1 year
  Number of falls

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle NICOLAS-VIRELIZIER, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fournier B, Nicolas-Virelizier E, Russo C, Perol O, Millet GY, Maire A, Delrieu L, Michallet AS, Assaad S, Belhabri A, Gilis L, Guillermin Y, Lebras L, Rey P, Santana C, Pretet-Flamand E, Terret C, Michallet M, Fervers B. Individualised physical activity programme in patients over 65 years with haematological malignancies (OCAPI): protocol for a single-arm feasibility trial. BMJ Open. 2021 Jun 3;11(6):e046409. doi: 10.1136/bmjopen-2020-046409. PMID 34083339